CLINICAL TRIAL: NCT04309019
Title: Constipation, Gut Microbiome, and Microbial-derived Uremic Toxins From the Gut Microbiota in HD Patients Is There a Relationship Between Them ?
Brief Title: Constipation, Gut Microbiome, and Microbial-derived Uremic Toxins From the Gut Microbiota in HD Patients
Status: Completed | Type: Observational
Sponsor: Tungs' Taichung Metroharbour Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 108080
Record Dates: First submitted 2020-03-11; First posted 2020-03-16 (Actual); Last update posted 2022-04-29 (Actual); Status verified 2022-04

CONDITIONS: Constipation; Inflammation
Keywords: constipation, , ,; gut microbiome; uremic toxins; inflammation
MeSH Terms: conditions — Constipation; Inflammation

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Chronic constipation is a prevalent, multifactorial gastrointestinal disorder, and its etiology and pathophysiology remain poorly understood. Recently studies using 16S rDNA-based microbiota profiling have demonstrated dysbiosis of gut microbiota in chronic constipation. In addition, alterations of fecal flora of the a group of severely constipated patients had been reported. Constipation, an indicator of gut dysbiosis in dialysis patients, may also pose a greater burden in dialysis patients. Some recent findings highlight the plausible link between the gut and the kidneys and provide additional insights into the pathogenesis of kidney disease progression and development of cardiovascular disease. Yet, the constipation in dialysis patients is usually ignored and not even draw the attention of dialysis physician as an ominous risk factor of constipated dialysis patients. In view of multiple factors link the gut and cardiorenal pathophysiology, and the scarcity of literature on this issue, the aim of this study is want to know if constipation can result in any changes to the intestinal microbiota and is it associated with inflammation, atherogenic profile and levels of microbial derived uremic toxins. Here, the investigators use both self-reported Bristol stool form scale (BSFS) scores and Roman IV criteria to diagnose constipation and 16S rDNA Illumina amplicon profiles of faecal samples of 90 dialysis patients to assess potential associations between microbiota composition and constipation. The relationship between uremic toxins and inflammation will also be explored in the dialysis suffering from constipation.

DETAILED DESCRIPTION:
Study Design and Population

Patients and Methods

This study will include 90 dialysis patients. Patients over age 20 years old and undergoing HD for at least 6 months will be enrolled. Patients with inflammatory diseases, cancer, AIDS, autoimmune disease, use of a central catheter for hemodialysis access, amputated limbs, pregnancy, and patients using catabolic drugs, antioxidant vitamin supplements pre, pro and symbiotic and antibiotics in the last 3 months before the start of this study were excluded. Dialysis duration was 4 hours per session, three times per week, with a blood flow >250 mL/min and a dialysate flow of 500 mL/min.

Analytic Procedures and Sample Processing

Blood samples will be drawn from each subject in the morning, after overnight fasting (for HD patients before a regular HD session). Plasma was separated (15 minutes, 30003 g, 4 C) and stored in -80 C until analysis.

Total concentrations of uremic toxins indoxyl sulfate(IS), p-cresol sulfate(PCS), and indoleacetic acid( IAA) are quantified by high-performance liquid chromatography (HPLC) with fluorescent detection.. Briefly, for binding competition, 200μl serum to which we added 20μl 0.50mM 1-naphthalenesulfonic acid (internal standard) was vortex-mixed with 250μl 0.24M sodium octanoate (binding competitor).After incubation at room temperature for 5min, we added 2ml cold acetone to precipitate proteins. Following vortex-mixing and centrifuging at 4 ◦C, 1860×g for 20 min, the supernatant was transferred to 12mm×100mm, GL 14 glass test tubes and 2ml dichloromethane was added. After vortex-mixing and centrifuging at 4 ◦C, 1860×g for 10min, 200μl of the upper layer was transferred to glass autosampler vials, followed by addition of 20μl 1M HCl and 15μl was injected onto the HPLC. The HPLC analysis was performed on an Agilent 1100 series LC (Santa Clara, CA),and Agilent ChemStations software were used for the chromatographic analysis. The separation was carried out on a ZORBAX SB-C18 Solv Saver Plus HPLC column (5 μm, 3.0 mm×150 mm).at a flow rate of 0.6 ml/min. Mobile phase A is 0.2% trifluoroacetic acid in Milli-Q water and mobile phase B is 0.2% trifluoroacetic acid in acetonitrile. The analytical method consists of an isocratic run with 92% mobile phase A for 23 min.. Each analytical run was followed by a 1.3 min washout gradient to 100% B. Column temperature was 25 ◦C, and autosampler tray temperature was 6 ◦C. We quantified the analytes by using the analyte to standard peak area ratio on a Agilent 1100 High Performance Fluorescence detector G1321A and Agilent 1100 Series UV-Visible detectors G1314A. Detector settings were λex 260 nm/λem288nm for p-cresyl sulfate and λex 280 nm/λem 390nm for indoxyl sulfate and IAA.

Total antioxidant activity (TAA) is measured in plasma using the Antioxidant Status Assay Kit (Calbiochem, Darmstadt, Germany) according to the manufacturer's protocol. The assay is defined as the ability of antioxidants in the plasma samples to prevent oxidation of 2,2'-azino-bis-(3-ethylbenz-thiazoline-6-sulfonic acid) (ABTS) by metmyoglobin. The amount of ABTS+ produced is monitored by reading the absorbance at 600 nm. The inter- and intra-assay coefficients of variation are 5.0% and 4.3%, respectively.

High-sensitivity protein C reactive (CRP), interleukin- 6 (IL-6), MCP-1, and Calprotectin were analyzed by immunoenzymatic assay (ELISA; R&D systems ). Routine laboratory parameters were measured by standard techniques.

Laboratory measurements

Total Antioxidant Status (TAS) kits purchased from Randox Laboratories Ltd. (Crumlin, UK) are applied for the assessment of the overall serum antioxidant capacity. It is based on the suppression of the formation of 2,2'-azinobis (3-ethylbenzothiazoline-6-sulfonate; ABTS*+), mediated mainly by the subsequent antioxidants: uric acid, protein thiol groups, ascorbic acid, and tocopherol. The plasma levels of MCP-1, IL-6, CRP, IL-17A and calprotectin are tested by commercially available human ELISA kit respectively, according to the manufacturer's instruction.

Stool DNA Isolation and 16S rDNA Gene Amplicon Sequencing

QI Aamp DNA Stool Mini Kit (51504; Qiagen, Germantown, MD) is used to extract gDNA from freshly collected feces samples from both mouse strains. The 16S rDNA gene variable regions V3-V6 are amplified by PCR using fecal gDNA. PCR comprised two consecutive steps. Primers targeting the 16S rDNA gene (italic) and specific primers carrying the 59M13/rM13 adapters (bold) 338FM13 (GTAAACGACGGCCAGTGCTCCTACGGGWGGCAGCAGT) and 1044R-rM13 (GGAAACAGCTATGACCATGACTACGCGCTGACGACARCCATG) are used to amplify the V3-V6 region of the bacterial 16S rDNA gene. After purification of PCR products using the NucleoSpin Gel and PCR Clean-Up Kit per the manufacturer's instructions, concentration and quality of the purified PCR products are assessed. To barcode each PCR product with a specific MID sequence and add the 454-specific Lib-L tag, a second PCR was performed using M13/rM13-specific primers containing the 454-specific Lib-L primers (underlined) A-M13 (CCATCTCATCCCTGCGTGTCTCCGACTCAG / MIDsequence/GTAAACGACGGCCAGG) and B-rM13 (CCTATCCCCTGTGTGCCTTGGCAGTCTCAGGGAAACAGCTATGA CCATGA).

Amplicons of the second PCR were pooled and purified by ethanol precipitation. Purified PCR products are run on a 0.8% agarose gel, bands corresponding to the barcoded 16S rDNA gene sequences are excised, and DNA was extracted using the NucleoSpin Gel and PCR Clean-Up Kit. DNA is eluted in ddH2O, further purified using AMPure Beads (Beckman Coulter, Inc., Brea, CA), and finally, resuspended in ddH2O. Concentration and quality of the purified barcoded sequences are assessed using a Nanodrop (Peqlab Biotechnology). Samples are stored at 220°C. Amplicon sequencing is performed at Eurofins on a 454 GS FLX Titanium Platform from one side (Lib-L-A) according to the recommended procedures for 454 Roche (Roche, Basel, Switzerland).

ELIGIBILITY:
Inclusion Criteria:

* Patients over age 20 years old
* Undergoing hemodialysis (HD) for at least 6 months

Exclusion Criteria:

* Inflammatory diseases
* Cancer
* AIDS
* Autoimmune disease
* Use of a central catheter for hemodialysis access
* Amputated limbs
* Pregnancy
* Using catabolic drugs
* Using antioxidant vitamin supplements
* Using symbiotic and antibiotics

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients have to be at least 20-years-old and and undergoing hemodialysis (HD) for at least 6 months.
Sampling Method: Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2020-03-10 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Serum uremic toxins such as indoxyl sulfate, p-cresol and IAA analysis | 1 years
  gut microbiota composition have been associated with increased production of indoxyl sulfate and p-cresyl sulfate, which is directly associated with endothelial dysfunction, inflammation and oxidative stress, and increases in the incidence of CVD and mortality.

SECONDARY OUTCOMES:
Stool DNA Isolation and 16S rDNA Gene Amplicon Sequencing | 1 years
  16S rDNA Illumina amplicon profiles of faecal samples to assess potential associations between microbiota composition and constipation.

CONTACTS AND LOCATIONS:
Overall Officials: Paik Seong Lim, PhD, Principal Investigator — Tungs' Taichung Metroharbour Hospital
Locations (1):
- Tungs' Taichung MetroHarbour Hospital, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided